CLINICAL TRIAL: NCT01048424
Title: Slow Paced-Respiration Intervention to Reduce Incontinence Trial (SPIRIT)
Acronym: SPIRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Alison Huang, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPIRIT001
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-10

CONDITIONS: Urinary Incontinence, Urge
Keywords: Urinary incontinence; Paced respiration
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paced respiration (Experimental): Participants will be instructed to practice slow-paced respiration for 15 minutes a day using the RESPeRATE device, and will also be given a Urinary Incontinence pamphlet containing general information about urinary incontinence and behavioral strategies for managing incontinence symptoms.
  Interventions: Device: RESPeRATE; Other: Urinary Incontinence Pamphlet
- Control (Placebo Comparator): Participants will be given a Urinary Incontinence pamphlet including general information about urinary incontinence and behavioral strategies for managing incontinence symptoms.
  Interventions: Other: Urinary Incontinence Pamphlet

INTERVENTIONS:
Device: RESPeRATE — RESPeRATE is a commercially available, "walkman-like" device manufactured by Intercure, Ltd. that measures chest/abdominal excursion during respiration using an elastic belt with a sensor placed around the torso over clothing. The device senses respiration and uses musical tones keyed to inhalation and exhalation to help the user slow respiration and prolong exhalation to a recommended goal of less than 10 breaths per minute. RESPeRATE is approved by the FDA for treatment of mild hypertension and has also been shown to decrease self-reported anxiety and stress, oxygen consumption, and respiratory rate.
  Arms: Paced respiration
Other: Urinary Incontinence Pamphlet — The urinary incontinence pamphlet will provide information about classification, pathophysiology, and management of urinary incontinence, including management strategies such as timed urination and pelvic muscle exercises.

SUMMARY:
Urgency incontinence is a common and burdensome problem in women. Current treatments for this condition, while effective, are associated with potentially disabling side effects and high rates of discontinuation. There is an urgent need for alternate treatments for urgency incontinence that are both clinically effective and well-tolerated by women in the community.

RESPeRATE is a commercially available "walkman-like" device that measures chest/abdominal excursion during respiration using an elastic belt with a sensor placed around the torso over clothing. The device senses respiration and uses musical tones keyed to inhalation and exhalation to help the user slow respiration and prolong exhalation to a recommended goal of less than 10 breaths per minute. RESPeRATE is approved by the US Food and Drug Administration (FDA) for treatment of mild hypertension, and use of the device has also been shown to decrease self-reported anxiety and stress, oxygen consumption, and respiratory rate. Because anxiety and stress are strongly associated with urgency incontinence, and common behavioral strategies for managing incontinence emphasize relaxation and slow breathing at the time of an urgency episode, paced respiration may also be useful in treating urgency incontinence and/or decreasing its burden on quality of life.

We propose to conduct a 6-week pilot randomized controlled trial of slow paced respiration using the RESPeRATE device among 30 women with urgency incontinence to assess the feasibility of recruiting and teaching women to use the RESPeRATE device as well as to gather preliminary data on the efficacy of slow paced respiration for treatment of urgency incontinence and related symptoms. Participants will complete a 7-day voiding diary and complete questionnaires to measure outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older who report urinary incontinence for greater than or equal to 3 months prior to screening
* Report that the majority of their incontinence episodes are associated with a sensation of urgency
* Record at least 7 urgency incontinence episodes per week on a screening 7-day voiding diary
* Able to walk to the toilet and use the toilet by themselves without difficulty
* Willing to refrain from initiating treatments that may affect their voiding pattern during the trial period
* Capable of understanding study procedures and giving informed consent

Exclusion Criteria:

* Current use of medical therapy for incontinence or use within the previous month (participants may be able to stop use of therapy and re-present for study)
* Currently pregnant, gave birth within the past 3 months, or planning pregnancy during the study period (approximately 2 months)
* Current urinary tract infection (screening dipstick urinalysis with leukocyte estrace, nitrites or blood) or a history or 4 or more urinary tract infections in the preceding year
* Report history of neurologic conditions such as stroke, multiple sclerosis, spinal cord injury, Parkinson's disease
* Report history of interstitial cystitis, fistula or hole in bladder or rectum, or birth defect leading to urine leakage
* Report history of pulmonary disease including emphysema, chronic bronchitis, or chronic obstructive pulmonary disease
* Measured resting blood pressure (average of 2 measures) less than 100/60 at screening or baseline examination
* Report any history of prior anti-incontinence or urethral surgery, pelvic cancer, or pelvic irradiation for any reason
* Report use of bladder botox, electrostimulation, bladder training, or pelvic floor exercise training (with certified practitioners) in the past 3 months
* Report other surgery to the pelvis (hysterectomy, oophorectomy, vaginal surgery, bladder surgery, colon surgery) during the past 3 months
* Report conditions that, in the judgment of the clinical center Principal Investigator, render potential participants unlikely to follow the protocol, including plans to move, substance abuse, significant psychiatric problems, or dementia
* Participation in another research study that involves investigational drugs or devices that could potentially confound the results of this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Huang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF-Mt. Zion Women's Health Clinical Research Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paced Respiration: Participants will be instructed to practice slow-paced respiration for 15 minutes a day using the RESPeRATE device, and will also be given a pamphlet containing general information about urinary incontinence and behavioral strategies for managing incontinence symptoms.
- Usual Care: Participants will be given a pamphlet including general information about urinary incontinence and behavioral strategies for managing incontinence symptoms.
Period: Overall Study
Arm/Group | Paced Respiration | Usual Care
Started | 10 | 10
Completed | 8 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paced Respiration | Usual Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 2 | 4 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 56.7 (10.9) | 54.73 (16.8) | 56 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Urgency Urinary Incontinence Episodes Per Week
Description: The number of incontinence episodes per week was calculated only over a 1-week period before the 6-week visit. There were no other interim outcomes assessment timepoints.
Time Frame: baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Control: Participants will be given a pamphlet including general information about urinary incontinence and behavioral strategies for managing incontinence symptoms.
Arm/Group | Paced Respiration | Control
Number analyzed (Participants) | 8 | 10
Percent Change | -33 (40) | -6 (50)

2. Secondary Outcome: Percent Change in Any Urinary Incontinence Episodes Per Week
Description: as for outcome 1
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Paced Respiration | Usual Care
Number analyzed (Participants) | 8 | 10
Percent Change | -18 (40) | -2 (40)

3. Secondary Outcome: Percent Change in Daytime Voiding Frequency.
Description: as for outcome 1
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Paced Respiration | Usual Care
Number analyzed (Participants) | 8 | 10
Percent Change | -9 (20) | 3 (30)

4. Secondary Outcome: Change in Overactive Bladder Symptoms
Description: The Overactive Bladder Questionnaire (OAB-Q). 0- to 100-point scale. Higher scores on the OAB-Q indicate greater bothersomeness and impact of overactive bladder symptoms.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paced Respiration | Usual Care
Number analyzed (Participants) | 8 | 10
Score on a Scale | -.63 (0.9) | -.44 (0.8)

5. Secondary Outcome: Change in Anxiety Symptoms
Description: Hospital Anxiety and Depression Scale. Anxiety Subscale range from 0 to 21, with scores of less than 8 indicative of absence of anxiety symptoms, 8 or above suggesting anxiety symptoms, and 12 or above suggesting generalized anxiety disorder.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paced Respiration | Usual Care
Number analyzed (Participants) | 8 | 10
Score on a Scale | -.78 (2.4) | -.57 (4.6)

6. Secondary Outcome: Change in Depression Symptoms
Description: Beck Depression Inventory. Range of 0-63 (0-9 normal; 10-16 mild; 17-29 moderate; 30-63 severe).
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paced Respiration | Usual Care
Number analyzed (Participants) | 8 | 10
Score on a Scale | -2.67 (3.7) | 2.25 (4.3)

7. Secondary Outcome: Change in Perceived Stress
Description: Cohen Perceived Stress Scale. Scores are scaled from 0 to 40, with higher scores indicated greater perceived stress.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paced Respiration | Usual Care
Number analyzed (Participants) | 8 | 10
Score on a Scale | -1.13 (3.5) | 4.13 (7.2)

8. Secondary Outcome: Change in Sleep Quality
Description: The Pittsburgh Sleep Quality Index. A global sleep quality score derived from the PSQI can be used to index overall quality of sleep over the prior one-week period. Global sleep quality scores are continuous (range 0-21), with high scores reflecting poor sleep quality.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paced Respiration | Usual Care
Number analyzed (Participants) | 8 | 10
Score on a Scale | -1.43 (2.0) | -.38 (2.4)

9. Secondary Outcome: Change in Incontinence- or Bladder-specific Quality of Life
Description: Incontinence Impact Questionnaire. Scores on the overall IIQ range from 0 to 400, with higher scores indicating greater overall impact on quality of life.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Paced Respiration | Usual Care
Number analyzed (Participants) | 8 | 10
Score on a Scale | -.15 (0.5) | -.06 (0.7)

ADVERSE EVENTS:
Arm/Group | Paced Respiration | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 1/8 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Paced Respiration (N=8) | Usual Care (N=10)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1/8 (1)
Cough (Infections and infestations) | 1 (1) | 2/8 (2)
Headache Issues (Nervous system disorders) | 0 (0) | 1/8 (1)
Increased Fatigue Issues (General disorders) | 1 (1) | 0/8 (0)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3/8 (3)
Light-Headedness Issues (Nervous system disorders) | 1 (1) | 0/8 (0)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1/8 (1)
Rapid Heart Beat Issues (Investigations) | 1 (1) | 0/8 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1/8 (1)
Swelling of both feet (General disorders) | 0 (0) | 1/8 (1)
Urinary Tract Infection (Investigations) | 1 (1) | 0/8 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes